CLINICAL TRIAL: NCT05865184
Title: Feasibility of Home-based, Ambient Passive Sensor Technology to Provide Early Warning of Health Decompensation by Detecting Deviations in Activities of Daily Living (ADLs) of Elderly Subjects With Diagnosed Chronic Disease
Brief Title: Evaluation of Home-based Sensor System to Detect Health Decompensation in Elderly Patients With History of CHF or COPD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sensorum Health Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Sensorum P-001
Record Dates: First submitted 2023-05-03; First posted 2023-05-18 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: COPD; Chronic Obstructive Pulmonary Disease; COPD Exacerbation; CHF; Congestive Heart Failure
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Heart Failure | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Passive monitoring: No intervention
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Data collection of clinically relevant signals using home-based sensor system

SUMMARY:
Sensorum Health (Sensorum) is conducting a pilot study to determine if Sensorum's proprietary passive sensor network can be used to identify signals of early health decompensation in subjects prior to a hospitalization for chronic disease exacerbation or other ambulatory care sensitive conditions. Successful early detection would provide a window of opportunity to intervene outside of the acute setting in future interventional studies.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 years or older
* Able to consent
* Documented history of diagnosis of chronic obstructive pulmonary disease (COPD) and/or congestive heart failure (CHF)
* Currently admitted to JSUMC for observation or as an inpatient with any diagnosis ≥1 prior hospital utilization events with any diagnosis (inpatient admissions, facility observation stays, or ED visits) in the past 12 months

Exclusion Criteria:

* Significant cardiac valvular disease
* End-Stage Renal Disease (ESRD)
* End-Stage CHF
* End-Stage COPD

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients admitted as inpatient to Jersey Shore University Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-09-28 (Actual); Primary Completion 2024-06-06 (Estimated); Study Completion 2024-06-06 (Estimated)

PRIMARY OUTCOMES:
Recall of AI in passive sensor system | 90 days
  Evaluation of AI ability to prospectively detect hospital utilization event
Precision of AI in passive sensor system | 90 days
  Evaluation of AI ability to precisely predict hospital utilization event

SECONDARY OUTCOMES:
Recall of sensor data review by trained nurses | 90 days
  Evaluation of nurse ability to prospectively detect hospital utilization event
Precision of sensor data review by trained nurses | 90 days
  Evaluation of nurse ability to precisely predict hospital utilization event

CONTACTS AND LOCATIONS:
Overall Officials: Swapnel Patel, MD, Principal Investigator — Jersey Shore University Medical Center, Hackensack Meridian Health
Locations (1):
- Jersey Shore University Medical Center, Hackensack Meridian Health, Neptune City, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No